CLINICAL TRIAL: NCT00731185
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Study on Efficacy and Safety of Mometasone Furoate Nasal Spray (MFNS) in the Post Surgical Treatment of Nasal Polyposis
Brief Title: Mometasone Furoate Nasal Spray for Treatment of Nasal Polyposis After Surgery (Study P03218)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P03218
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Nasal Polyps
Keywords: functional; endoscopic; sinus; surgery
MeSH Terms: conditions — Nasal Polyps; Fistula | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mometasone Furoate Nasal Spray (MFNS) (Experimental): MFNS 200 mcg (2 sprays of 50 mcg in each nostril) once daily in the morning
  Interventions: Drug: Mometasone Furoate Nasal Spray
- Placebo (Placebo Comparator): Placebo nasal spray (2 sprays of 50 mcg in each nostril) once daily in the morning
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone Furoate Nasal Spray — MFNS 200 mcg (2 sprays of 50 mcg in each nostril) once daily in the morning for up to 24 weeks or until relapse
  Other Names: Nasonex; SCH 032088
  Arms: Mometasone Furoate Nasal Spray (MFNS)
Drug: Placebo
  Other Names: Placebo (2 sprays of 50 mcg in each nostril) once daily in the morning for up to 24 weeks or until relapse
  Arms: Placebo

SUMMARY:
This study was conducted to evaluate the effectiveness of mometasone nasal spray in preventing polyp relapse/symptom worsening in patients after surgical treatment of nasal polyps. Patients who met Screening eligibility underwent endoscopic sino-nasal surgery (FESS) on visit 2. Mometasone nasal spray or placebo was started about 2 weeks after surgery and continued for up to 24 weeks or until relapse.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Bilateral nasal polyps
* Fulfill criteria for polypectomy (be indicated for surgical - FESS - treatment)

Exclusion Criteria:

* Polypectomy within the last 6 months
* Unhealed nasal surgery/trauma
* >5 previous polypectomies
* Female of childbearing age who is pregnant, lactating, or not using active contraceptive methods
* Nasal infection
* Pulmonary tuberculosis
* Cystic fibrosis, glaucoma, clinically significant cardiovascular, pulmonary, renal, hepatic, metabolic, hematological, or neurological disease
* Immunocompromised
* Rhinitis medicamentosa (rebound congestion following misuse of nasal decongestants)
* Known hereditary mucociliary dysfunction
* Significant nasal structure abnormalities
* Asthmatic attack within the past 30 days
* Asthmatic patients requiring >1000 mcg beclomethasone or equivalent
* Asthmatic patients not stable on corticosteroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2003-09-01 (Actual); Primary Completion 2005-09-01 (Actual); Study Completion 2005-09-01 (Actual)

PRIMARY OUTCOMES:
Time to relapse in polyp score after surgery | Assessment for relapse was performed at every study visit (up to 24 weeks of treatment)

SECONDARY OUTCOMES:
Signs and symptom scores | All study visits (up to 24 weeks of treatment)
Quality of life, peak nasal inspiratory flow, olfaction threshold | Measured starting 1 week after treatment up to 24 weeks of treatment
Adverse events | Throughout the whole study after the Screening period.

REFERENCES:
- [Derived] Stjarne P, Olsson P, Alenius M. Use of mometasone furoate to prevent polyp relapse after endoscopic sinus surgery. Arch Otolaryngol Head Neck Surg. 2009 Mar;135(3):296-302. doi: 10.1001/archoto.2009.2. PMID 19289710